CLINICAL TRIAL: NCT05317104
Title: The Effect of Aerobic Exercise Training in Collegiate eSport Team Players on Reaction Time and Cognitive Functions- A Randomized, Single Blind, Controlled Trial
Brief Title: The Effect of Aerobic Exercise Training on Collegiate eSport Team Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Pelin Pişirici, Assistant Professor, PT, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Esport-05/03/2022
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Screen Time; Performance Enhancing; Injury Prevention; Executive Function; Cardiovascular Training
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 30 esports players aged 18-25, playing in the university esports team, will be included in the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All outcomes and measurements are done by a blinded assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Group (Experimental): Intervention group will be included in a program consisting of warm-up, loading and cool-down periods. Maximum Heart Rate (MHR) method will be used to determine the intensity of aerobic exercise training. Since moderate aerobic exercise training was aimed, exercise training will be given in 55-74% of MHRs. Exercise training will be started at mild-moderate intensity. Afterwards, within the limits that the person can tolerate and does not cause complications, with 5-10 minute increments every 1-2 weeks, the person will progress without muscle pain, injury, respiratory distress or fatigue due to overload. Polar H9 Heart Rate Sensor, which will be worn on the chest, will be used to monitor heart rate during exercise training.
  Aerobic exercise training will be given in accordance with the procedures determined on the treadmill in the laboratory environment, with a program consisting of 6-week.
  Interventions: Other: Aerobic exercise
- Control Group (No Intervention): No intervention will be made other than evaluations. However, in order for the participants in this group to achieve the same health gains, they will remain under follow-up and control to apply the same aerobic exercise training program after the study is completed.

INTERVENTIONS:
Other: Aerobic exercise — For 6 weeks, 3 times a week, aerobic exercise will be performed with a treadmill at 55-74% of the maximal heart rate.
  Arms: Aerobic Exercise Group

SUMMARY:
E-sports, which is called video games that are played in a competitive and organized way in a virtual environment, individually or in like teams, continues to increase its popularity by reaching individuals of all ages with the acceleration it has gained to worldwide.

The major keys to performance in e-sports, which include games in many different categories; tactical and cognitive abilities that depend on executive functions such as attention, perception, memory, and multitasking. It also requires play skills that include fluent and coordinated movements, such as hand-eye coordination. Therefore, the reaction time among the players plays a decisive role in the performance.

The sedentary life-induced physical, mental and spiritual health of the e-sports player who is in front of the screen for a long time is negatively affected, and it is seen that the accuracy in the executive functions of the athlete decreases and results in impulsivity. Physical activity can be considered as a good opportunity for performance, as physical, cognitive and spiritual improvements will contribute positively to the performance of the athlete. Aerobic exercise, which is widely performed today for physical activity, has positive effects on both physical, cognitive and psychosocial aspects.

This study was designed as a randomized controlled, single-blind, prospective study to examine the effect of aerobic exercise training on reaction time, neuropsychological parameters and mood in e-sports players playing in university e-sports team.

DETAILED DESCRIPTION:
E-sports, which are called video games that are played in a competitive and organized manner in a virtual environment, individually or in teams, in line with a certain goal, are taking place today based on the principle of directing virtual avatars. Following the increase in personal computer use, it continues to increase its popularity by reaching individuals of all ages, while gaining a worldwide popularity with players predominantly consisting of younger population.

The major keys to performance in e-sports, which include games in many different categories; Tactical and cognitive abilities that depend on executive functions such as attention, perception, memory, and multitasking. It also requires play skills that include fluent and coordinated movements, such as hand-eye coordination. Therefore, the reaction time among the players plays a decisive role in the performance.

Since the e-sports player, whose average career years are known to be short, will regularly train 5.5-10 hours a day in order to continue with maximum performance and improve their skills, many of the players earn a sedentary life by not participating in any physical activity. Although the increase in the time spent in front of the screen brings success, physical and mental health due to the sedentary life gained is negatively affected, and it is seen that the accuracy in executive functions decreases and results in impulsivity as it is continued without rest. In addition to these, it will be possible to say the presence of depression and anxiety.

According to the guidelines published by the World Health Organization, it has been observed that individuals aged 18-64 are recommended at least 150-300 minutes of moderate-intensity aerobic activities per week or at least 75-150 minutes of vigorous aerobic activities.

Physical activity can be considered as a good opportunity for performance, since the physical-cognitive system that works smoothly in e-sports players will contribute positively to the performance of the athlete. Since physical activity also contributes to mental healing, it is thought that the athlete's chance of success will be higher by causing a positive effect on the performance of the player.

Aerobic exercise, known as activities in which the major muscle groups of the body are moved rhythmically for a continuous period of time, increase synaptic plasticity, while aerobic exercise is known to improve attention and affect reaction times in direct proportion to attention. Positive effects of aerobic exercise are observed in psychosocial aspects as well as in cognitive development.

Reaction time; 3 separate tests, visual, auditory and audio-visual, will be evaluated with computer aided Microgate-Optojump Next measuring device. Neuropsychological evaluation; short-term memory, attention, information processing speed, and problem-solving skills will be evaluated with Corsi Block Task, Stroop Test, Wisconsin Card Sorting Test, Fitts Law Test and Digit Span Test. Mood evaluation will be done with Beck Depression Inventory and Beck Anxiety Inventory. Before people are included in the exercise training protocol, knowing the person's maximum exercise capacity will determine an effective program and the person/situation where we need to end the exercise, so aerobic exercise capacity will be done with the '20 Meter Shuttle Run Test', which is a maximal field test.

This study was designed as a randomized controlled, single-blind, prospective study to examine the effect of aerobic exercise training on reaction time, neuropsychological parameters and mood in e-sports players playing in university e-sports team.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-25
* Playing e-sports for at least 1 year
* Training at least 2 hours per a day
* Playing one of the types of games played using a computer
* Playing on a university esports team
* Volunteer

Exclusion Criteria:

* Being diagnosed with any neurological, psychiatric, cardiopulmonary, rheumatological, orthopedic and oncological disease
* Having a history of injuries involving the musculoskeletal system
* Having a congenital/acquired mental or physical disability that prevents participation in the study
* Using sleeping pills due to the sleep problem experienced
* Playing games with devices such as mobile phones, consoles
* Failure to complete exercise capacity measurement

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-25 (Actual)

PRIMARY OUTCOMES:
Reaction Time | Begining of the study, 6 weeks after the baseline
  Reaction Time: Reaction time; 3 separate tests, visual, auditory and audio-visual, will be evaluated with a computer-aided Microgate-Optojump measuring device. Evaluation; using a fixed chair, the athlete's feet should be made in full contact position on the floor.

SECONDARY OUTCOMES:
Corsi Block Task | Begining of the study, 6 weeks after the baseline
  The test aiming to measure visual-spatial short-term memory will be done on a digital platform. In the test, which starts with two blocks and increases in difficulty, the test will continue until nine blocks are completed correctly in the desired order. The test will automatically terminate if completed without errors or if repeated errors are made at the same level.
Stroop Test | Begining of the study, 6 weeks after the baseline
  Although there are different standardizations of the Stroop test, which is used as the gold standard in attention measurements, its two tasks will be tested. The participant will be tested with the tasks of reading the colored words and telling the color of the colored words. The test will be able to record the desired color with the correct data and will be measured by the elapsed time. The time difference between the two missions will give the score.
Wisconsin Card Sorting Test | Begining of the study, 6 weeks after the baseline
  The test used to evaluate cognitive flexibility will be done on a digital platform. Test; It is based on matching the response cards with the stimulus cards through the feedbacks (True/False) given by a series of cards with 4 different stimulus cards at each stage, and a total of 64 response cards, categorized by subject, color, shape and number types. After the card to be matched is shown, it is stated that the selected figure is only true or false, while it is not specified under which category the choice is desired. Test score criteria; The total obtained will include data such as error, number of trials, perseverative and non-perseverative data. The main purpose is to measure how well it adapts to changing rules.
Fitts Law Test: | Begining of the study, 6 weeks after the baseline
  The test, which aims to measure the speed of information processing, will be held on a digital platform. Maximum performance will be based on the ability to follow the constantly changing box with hand-eye coordination. In the test, the speed and accuracy of the movement will be calculated by the movement of the mouse cursor in the direction of the instructions given to the participants, and the time it takes to reach the shapes in the targeted sizes and intervals.
Digit Span Test | Begining of the study, 6 weeks after the baseline
  It will be done to measure attention and working memory. The main task of the test is to recall the data in the desired order. Only the Forward part of the test, which consists of two parts, will be done. After listening to the previously recorded data one by one, the participant will be expected to write it down on a piece of paper after each recording. The test will be terminated if wrong at the same level twice. The level reached will be the test score.
Beck Depression Inventory | Begining of the study, 6 weeks after the baseline
  A 21-item inventory will be used as an aid in quantitatively measuring the presence and intensity of depression symptoms. 0-9 points are interpreted as minimal, 10-16 points as mild, 17-29 points as moderate and 30-63 points as severe depression.
Beck Anxiety Inventory | Begining of the study, 6 weeks after the baseline
  The inventory created to differentiate anxiety from depression will be used to measure the level of anxiety. In the 21-item inventory, 0-7 points indicate the presence of minimal anxiety, 8-15 points mild, 16-25 points moderate and 26-63 points severe anxiety.
20 Meter Shuttle Run Test: | Begining of the study, 6 weeks after the baseline
  The '20 Meter Shuttle Run Test' will be used because knowing the person's maximum exercise capacity before being included in the exercise training protocol will determine the person/situation we need to end the exercise with. The test will be performed in accordance with the established procedures. The test will be terminated if it fails to cover the required path before the 'beep' stimulus twice, or if there is a desire to quit the test due to fatigue during the test. The number of shuttles and vital signs will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Beyza Çoban, PT, Principal Investigator — Bahçeşehir University, Graduate Education Institute, Physical Therapy and Rehabilitation; Sena Vargel, PhD (c), PT, Study Chair — Bahçeşehir University, Health Sciences Faculty, Physiotherapy and Rehabilitation; Selen Gür Özmen, MD, Associate Prof., Study Chair — Bahçeşehir University, Health Sciences Faculty, Physiotherapy and Rehabilitation; Pelin Pişirici, PhD, PT, Study Director — Bahçeşehir University, Health Sciences Faculty, Physiotherapy and Rehabilitation
Locations (1):
- Bahcesehir University, Istanbul, Besiktas, Turkey (Türkiye)